CLINICAL TRIAL: NCT04584151
Title: Does Bilateral Continuous Peri Operative Erector Spinae Plane (ESP) Block Improve the Enhanced Recovery Program After Liver Transplantation in Recipient Patient
Brief Title: Perioperative Analgesia by ESP Catheter on Recipient for Liver Transplantation
Acronym: ESPLIVERRec
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Surgeon left the team
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VINMEC LT REC
Record Dates: First submitted 2020-09-21; First posted 2020-10-12 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Liver Transplant Disorder

STUDY DESIGN:
Intervention Model Description: randomized controlled prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention): Peri operative analgesia by opioid
- Continuous regiona analgesia (Experimental): Peri operative algesia by continuous bilateral ESP catheters
  Interventions: Procedure: regional analgesia

INTERVENTIONS:
Procedure: regional analgesia — Insertion of bilateral ESP catheters
  Arms: Continuous regiona analgesia

SUMMARY:
Enhanced recovery after surgery (ERAS) programs were developed by Prof Henrik Kehlet in Denmark to reduce the hospitalization and improve the surgical outcomes. In these programs pain relief by regional analgesia techniques are highly recommended to reduced as much as possible the opioids used with their side effects. This program was created for colo-rectal surgeries and extended to other surgeries. In Liver transplants different programs has been described top reduce the use of peri-operative opioids but no with the ESP Animal and molecular studies in chronic pain showed the activation of glial cells, Monocytes and lymphocite K similar to the reaction during severe septis with immune reaction and toll like receptor activation. Regional anaesthesia analgesia is blocking this activation of Tool Like Receptors (TLR4) One of the discharge criteria after liver transplantation is the equilibrium of plasmatic cyclosporin Our hypothesis is with regional analgesia to avoid any immune disorder due to pain and reach earlier the discharge criteria than with standard analgesia Improve the quality of recovery and reduce the hospitalization stay after liver transplantation

DETAILED DESCRIPTION:
1. Goals:

   Compare quality of analgesia and quality of recovery between bilateral ESP bilateral catheters versus Opioid analgesia in adult included in an enhanced recovery program after liver transplantation Show that the addition of peri-operative regional analgesia improves the enhanced recovery program after open liver transplant in recipient patient .
2. Methodology:

   •Selection criteria: Age > 18 years old Have a clinical indication for Liver transplantation ( list for surgeries listed in full proposal) Agree to participate in the trial

   •Exclusion criteria: Use of chronic opioid Contra-indication tom perform ESP catheter (Infection near puncture point, Severe thoracic scoliosis, allergy to local anaesthetics) A diagnosis of a chronic pain condition Depression or other psychiatric diagnosis

   • Study design: Prospective Randomized Controlled Trial.

   Patients who agree to join the study will be randomized into 2 groups:

   Group 1 (Control group): standard of care in Liver donation : Intra operative analgesia by Opioid Sufentanil and post operative analgesia by Patient Controlled analgesia (PCA) opioid morphine Group 2 (treatment group): Standard peri-operative analgesia for Liver donation in our hospital since we use regional anaesthesia as first line treatment for peri operative analgesia Bilateral ESP catheters with continuous regional analgesia by infusion of local anaesthetic (Ropivacaine)

   Sample size: We expected to reduce the length of stay for liver receipt from 11 ± 2.22 days in ERAS group to 8 ± 2.22 days in the ESP group The sample size of 10 patients per group is required to detect such changes assuming a confidence interval of 95% with a power of 90% and alpha = 0.05. Considering 20% of drop-out, the total sample size is 40 patients (20 patients each group)
3. Project outcomes:

   * Primary outcomes Length of stay in Hospital Our estimation based on our previous studies for ESP and the literature for ERAS programs in open heart surgeries
   * Secondary outcomes Time to extubation Duration of stay in ICU Time to 1st mobilisation Opioid consumption in relation with VAS Rest and mobilization

Patient satisfaction:

* Quality of recovery scoring 15 items (QOR 15)
* Pain at 1 month rest and mobilization + Quality of Life scoring (QOL36)

ELIGIBILITY:
Inclusion Criteria:

* age clinical indication for liver transplantation agree to participate and signed consent

Exclusion Criteria:

* Use of chronic opioid contra indication to perform ESP cathters Diagnosis of a chronic pain condition except liver disease Psychiatric or depression disorder allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Length of stay in hospital | up to 30 day
  Time to reach the criteria of hospital discharge after liver transplantation

SECONDARY OUTCOMES:
Duration of stay in Intensive care Unit (ICU) | up to 72 hours
  Time to reach the criteria of ICU discharge after liver transplantation
Quality of recovery: score | up to 30 days
  Score on 15 criteria for quality of recovery from 0= very poor to 150 = excellent

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - VinMec INternational hospital, Hanoi
  - VinMec INternational hopspital, Hanoi

IPD SHARING:
Plan to Share IPD: No